CLINICAL TRIAL: NCT07003503
Title: Explore the Risk Factors for Antenatal Mental Disorders in Pregnant Women With Hyperglycemia
Status: Not yet recruiting | Type: Observational
Sponsor: Shenzhen Hospital of Southern Medical University (Other)
Responsible Party: Principal Investigator, Zonglian Guo, principle investigator, Shenzhen Hospital of Southern Medical University
Other Study IDs: NYSZYYEC2024K13OR001
Record Dates: First submitted 2025-04-22; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Hyperglycemia; Mental Disorder; Pregnancy Complications
Keywords: hyperglycemia; antenatal mental disorder; pregnancy complication
MeSH Terms: conditions — Hyperglycemia; Mental Disorders; Pregnancy Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pregnant women with hyperglycemia: Inclusion criteria: ① Pregnant women were confirmed as having gestational diabetes through biochemical examinations and glucose tolerance tests, etc. ② Possess the abilities of listening, speaking, reading, writing and comprehension, and be capable of effective communication; ③ Age: 18-45 years old (including 18 and 45 years old); ④ Informed consent and voluntary participation in the research; ⑤ Gestational age: 28 to 37 weeks (including 28 weeks but excluding 37 weeks).
  Exclusion criteria: ① Abnormal fetuses and multiple pregnancies; ② Other pregnancy complications and comorbidities, such as heart disease, preeclampsia, liver disease, etc. ③ There is a history of mental illness or mental disorders in the past. ④ Those who are unable to communicate effectively by using listening, speaking, reading and writing skills; ⑤ Patients with diabetes mellitus complicated with pregnancy; ⑥ Those who use psychotropic or neurotropic drugs.

SUMMARY:
This study aims to investigate the current situation and risk factors of adverse mental disorders in pregnant women with hyperglycemia. it could include any of the following: 18-45 years old pregnant women with hyperglycemia. The main question is to answer the risk factor for antenatal mental disorder. participants need to complete a self-report questionnaire.

DETAILED DESCRIPTION:
study design: This is a cohort study which will be conducted in the Shenzhen Hospital of Southern Medical University. Inclusion criteria: ① Pregnant women were confirmed as having gestational diabetes through biochemical examinations and glucose tolerance tests, etc. ② Possess the abilities of listening, speaking, reading, writing and comprehension, and be capable of effective communication; ③ Age: 18-45 years old (including 18 and 45 years old); ④ Informed consent and voluntary participation in the research; ⑤ Gestational age: 28 to 37 weeks (including 28 weeks but excluding 37 weeks).

Exclusion criteria: ① Abnormal fetuses and multiple pregnancies; ② Other pregnancy complications and comorbidities, such as heart disease, preeclampsia, liver disease, etc. ③ There is a history of mental illness or mental disorders in the past. ④ Those who are unable to communicate effectively by using listening, speaking, reading and writing skills; ⑤ Patients with diabetes mellitus complicated with pregnancy; ⑥ Those who use psychotropic or neurotropic drugs.

sample size: According to the sample size calculation formula of multivariate analysis, N=Zα/22×P(1-P)/δ2, P was 40.38% of the incidence of depression in pregnant women with gestational diabetes mellitus (GDM) as reported in the literature. When the test level α is set at 0.05, Zα/2=1.96; δ represents the allowable error, and δ=0.05. Therefore, the sample size obtained is 370 cases. Adding a 20% invalid questionnaire rate, the sample size obtained was 444 cases.

procedure: pregnant women who were diagnosis hyperglycemia through OGTT test between 24-28 gestational weeks will be enrolled in this study. When they were admitted to obstetric department when they had gestational week greater than 32 weeks to have childbirth, researchers will sent self-repot questionnaire to them after getting consent. The sequence of data collection is in the order of hospitalization time. A QR code will be gave them, when they tickle the join button which means they would like to participant this study. After getting consent from participants, researchers need to collect social demographic and mental health information from their electric medical record. Data processing was conducted using SPSS and R. Kolmogorov-smirnov was selected to detect whether continuous variables conform to the normal distribution. A P value <0.05 was considered statistically significant.

General information: Categorical variables are represented by frequency and percentage (%); For continuous variables, if they conform to a normal distribution, the mean ± standard deviation (x±SD) is used; otherwise, the median and interquartile range (M, IQR) are used.

LASSO regression analysis: LASSO regression analysis was conducted based on the questionnaire results of the modeling group. Taking whether adverse psychology occurred as the dependent variable and the questionnaire items of risk factors for adverse psychology in pregnant women with gestational diabetes mellitus (GDM) as independent variables, R was used to preliminarily screen the risk factors through tenfold cross-validation of LASSO regression.

Binary Logistic regression analysis: Taking the occurrence of adverse psychology as the dependent variable and the risk factors initially screened out by LASSO regression analysis as the independent variables (with independent variable assignment), binary Logistic regression analysis was conducted on the data of the modeling group. The Hosmer-Lemeshow test was conducted for goodness-of-fit examination. A p > 0.05 indicated a good fit of the model. Collinearity test: The variance inflation factor (VIF) is used for the collinearity test to detect the degree of correlation among the independent variables. A VIF > 10 indicates a strong collinearity.

Quality control Train data collectors to accurately assess the usage methods of the tools; After the data is collected and organized, it is checked and entered by two people to ensure the accuracy of the data.

③ Data analysis was conducted by two independent researchers. In case of any discrepancy, it was verified by a third independent researcher.

ELIGIBILITY:
Inclusion Criteria:

* The pregnant woman was confirmed to have gestational diabetes through biochemical tests and glucose tolerance tests, etc.
* Possess the abilities of listening, speaking, reading, writing and comprehension, and be capable of effective communication;
* Age: 18-45 years old (including 18 and 45 years old);
* informed consent and voluntary participation in the research;
* Gestational age: 28 to 37 weeks (including 28 weeks but excluding 37 weeks).

Exclusion Criteria:

* Abnormal fetuses, multiple pregnancies;
* Other pregnancy complications and comorbidities, such as heart disease, preeclampsia, liver disease, etc.
* There is a history of mental illness or mental disorders in the past.
* Those who are unable to communicate effectively by using listening, speaking, reading and writing skills;
* Patients with diabetes mellitus complicated with pregnancy;
* Those who use psychotropic or neurotropic drugs.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants should follow inclusive and exclusive criteria.
Sampling Method: Non-Probability Sample
Enrollment: 635 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
patient health questionnaire -9 (PHQ-9) score | Participants were administered in the hospital to deliver the baby.
  In the first, second and third trimesters, due to the government's policy, all pregnancies need to complete a EDSS if they want. When the pregnancies were diagnosed with hyperglycemia, a consent form was sent to them. After getting consent from them, researchers will retrospectively collect their medical records and EDSS scores in the government system when the participants were administrated in hospital to deliver the baby.
  the interpretation of PHQ-9: Total scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe and severe depression, respectively.

SECONDARY OUTCOMES:
Generalized Anxiety Disorder-7 scale score (GAD-7) | Participants were administered in the hospital to deliver the baby.
  In the first, second and third trimesters, due to the government's policy, all pregnancies need to complete a GAD-7 if they want. When the pregnancies were diagnosed with hyperglycemia, a consent form was sent to them. After getting consent from them, researchers will retrospectively collect their medical records and EDSS scores in the government system when the participants were administrated in hospital to deliver the baby.
  interpretation for GAD-7: It's a self-administered questionnaire with 7 questions, each scored from 0 to 3, totaling a possible score of 21. Scores of 5, 10, and 15 are often used as cut-offs to indicate mild, moderate, and severe anxiety, respectively.

IPD SHARING:
Plan to Share IPD: Yes
protocol
Supporting Information: Study Protocol

REFERENCES:
- [Background] Delanerolle G, Phiri P, Zeng Y, Marston K, Tempest N, Busuulwa P, Shetty A, Goodison W, Muniraman H, Duffy G, Elliot K, Maclean A, Majumder K, Hirsch M, Rathod S, Raymont V, Shi JQ, Hapangama DK. A systematic review and meta-analysis of gestational diabetes mellitus and mental health among BAME populations. EClinicalMedicine. 2021 Jul 14;38:101016. doi: 10.1016/j.eclinm.2021.101016. eCollection 2021 Aug. PMID 34308317
- [Background] DOI:10.16766/j.cnki.issn.1674-4152.003467.
- [Background] Thiele GA, Ryan DM, Oberlander TF, Hanley GE. Preconception mental health and the relationship between antenatal depression or anxiety and gestational diabetes mellitus: a population-based cohort study. BMC Pregnancy Childbirth. 2022 Aug 31;22(1):670. doi: 10.1186/s12884-022-05002-5. PMID 36045319
- [Background] Schmitt A, Bendig E, Baumeister H, Hermanns N, Kulzer B. Associations of depression and diabetes distress with self-management behavior and glycemic control. Health Psychol. 2021 Feb;40(2):113-124. doi: 10.1037/hea0001037. Epub 2020 Nov 30. PMID 33252963
- [Background] Riggin L. Association Between Gestational Diabetes and Mental Illness. Can J Diabetes. 2020 Aug;44(6):566-571.e3. doi: 10.1016/j.jcjd.2020.06.014. Epub 2020 Jun 22. PMID 32792108
- [Background] https://www.mdpi.com/1660-4601/17/11/3767.
- [Background] Mazumder T, Akter E, Rahman SM, Islam MT, Talukder MR. Prevalence and Risk Factors of Gestational Diabetes Mellitus in Bangladesh: Findings from Demographic Health Survey 2017-2018. Int J Environ Res Public Health. 2022 Feb 23;19(5):2583. doi: 10.3390/ijerph19052583. PMID 35270274
- [Background] Ye W, Luo C, Huang J, Li C, Liu Z, Liu F. Gestational diabetes mellitus and adverse pregnancy outcomes: systematic review and meta-analysis. BMJ. 2022 May 25;377:e067946. doi: 10.1136/bmj-2021-067946. PMID 35613728